CLINICAL TRIAL: NCT06378944
Title: INDOCYANINE GREEN for SELECTIVE SENTINELLA AXILLARY LYMPH NODE BIOPSY in PATIENTS with BREAST CANCER
Brief Title: Selective Sentinella Lymph Node Biopsy with Indocyanine Green in Patients with Breast Cancer
Acronym: INSEAN
Status: Recruiting | Type: Observational
Sponsor: Omphis Foundation (Other)
Responsible Party: Principal Investigator, Sandra Lopez Gordo, Doctor and head of the department of breast cancer unit Sandra Lopez Gordo, Omphis Foundation
Other Study IDs: 61/23
Record Dates: First submitted 2024-04-01; First posted 2024-04-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: lymph node detection; indocyanine green; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Technetium-99

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Application of green indocyanine colorant — The day of the surgery 1 ml of green indocyanine colorant will be applicated periareolar. After 5 minutes the lymph node will be detected and extracted
Drug: Technetium99 — Application of a periareolar injectionof TEchnetium 99 in order to detect the axillary lymph node

SUMMARY:
The current observational study aims to perform the sentinel lymph node in breast cancer in the usual way with technetium 99 and add a second tracer, indocyanine green. The objective is to evaluate the detection rate of the lymph node with indocyanine green compared to the usual technique.

DETAILED DESCRIPTION:
In the operating room 1 ml of indocyaninge grenn will be injectec periareolar . After 5 minutes the lymph node will be detected and extracted. The comparison between the lymph nodes detected with Technetium 99 and indocyanine green will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age with breast cancer who are candidates for sentinel lymph node detection will be included.
* N0 patients or patients who have undergone target axillary detection with good response

Exclusion Criteria:

* Lymphadenectomy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with breast cancer who recieve surgery and required to perform lymph node detection
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Sentinel lymph node detected. Scale of numbers | patients included from 1 January of 2024 til January 1 2029
  Number of lymph node detected with Indocyanine green and number of lymph node detected iwth techetium 99. Scale of numbers

SECONDARY OUTCOMES:
Number of possitive lymph nodes | patients included from 1 January of 2024 til January 1 2029
  assess whether there are differences in affected lymph nodes detected with indocyanine green or technetium 99 Number of possitive lymph nodes iwh indocyanine green and with technetium 99
surgery time in minutes | patients included from 1 January of 2024 til January 1 2029
  Time in minutes from skin incision to lymp node removal.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lopez gordo, Study Director — 46873584K
Locations (1):
- Sandra Lopez Gordo, Cerdanyola del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krag DN, Weaver DL, Alex JC, Fairbank JT. Surgical resection and radiolocalization of the sentinel lymph node in breast cancer using a gamma probe. Surg Oncol. 1993 Dec;2(6):335-9; discussion 340. doi: 10.1016/0960-7404(93)90064-6. PMID 8130940
- [Background] Giuliano AE, Kirgan DM, Guenther JM, Morton DL. Lymphatic mapping and sentinel lymphadenectomy for breast cancer. Ann Surg. 1994 Sep;220(3):391-8; discussion 398-401. doi: 10.1097/00000658-199409000-00015. PMID 8092905
- [Background] Goyal A, Newcombe RG, Chhabra A, Mansel RE; ALMANAC Trialists Group. Factors affecting failed localisation and false-negative rates of sentinel node biopsy in breast cancer--results of the ALMANAC validation phase. Breast Cancer Res Treat. 2006 Sep;99(2):203-8. doi: 10.1007/s10549-006-9192-1. Epub 2006 Mar 16. PMID 16541308
- [Background] Kitai T, Inomoto T, Miwa M, Shikayama T. Fluorescence navigation with indocyanine green for detecting sentinel lymph nodes in breast cancer. Breast Cancer. 2005;12(3):211-5. doi: 10.2325/jbcs.12.211. PMID 16110291
- [Background] Jeremiasse B, van den Bosch CH, Wijnen MWHA, Terwisscha van Scheltinga CEJ, Fiocco MF, van der Steeg AFW. Systematic review and meta-analysis concerning near-infrared imaging with fluorescent agents to identify the sentinel lymph node in oncology patients. Eur J Surg Oncol. 2020 Nov;46(11):2011-2022. doi: 10.1016/j.ejso.2020.07.012. Epub 2020 Aug 3. PMID 32826112
- [Background] Goonawardena J, Yong C, Law M. Use of indocyanine green fluorescence compared to radioisotope for sentinel lymph node biopsy in early-stage breast cancer: systematic review and meta-analysis. Am J Surg. 2020 Sep;220(3):665-676. doi: 10.1016/j.amjsurg.2020.02.001. Epub 2020 Feb 7. PMID 32115177
- [Background] Kedrzycki MS, Leiloglou M, Ashrafian H, Jiwa N, Thiruchelvam PTR, Elson DS, Leff DR. Meta-analysis Comparing Fluorescence Imaging with Radioisotope and Blue Dye-Guided Sentinel Node Identification for Breast Cancer Surgery. Ann Surg Oncol. 2021 Jul;28(7):3738-3748. doi: 10.1245/s10434-020-09288-7. Epub 2020 Nov 6. PMID 33156466